CLINICAL TRIAL: NCT01772641
Title: A Combination of Scheduled Reduced Smoking With Varenicline to Enhance Cessation
Brief Title: A Smoking Intervention Study Using Scheduled Gradual Reduction With Varenicline to Help With Cessation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty recruiting and retaining participants
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joel Erblich, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 10-0879; 5R34DA031327-02 (NIH)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Nicotine Addiction
Keywords: cigarette; smoking; cessation; varenicline; scheduled reduction; craving
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Scheduled Gradual Reduction + Varenicline (Experimental): Participants will be given the behavioral intervention of Scheduled Gradual Reduction along with the smoking cessation drug, Varenicline.
  Interventions: Other: Scheduled Gradual Reduction + Varenicline
- Scheduled Gradual Reduction + Placebo Drug (Experimental): Participants will be given the behavioral intervention, SGR, along with a placebo drug matching the schedule of the VN group.
  Interventions: Other: Scheduled Gradual Reduction + Placebo Drug
- Basic Advice + Varenicline (Experimental): Participants will be given basic advice about quitting smoking along with the smoking cessation drug Varenicline
  Interventions: Other: Basic Advice + Varenicline
- Basic Advice + Placebo Drug (Placebo Comparator): Participants will be given basic advice along with a placebo drug matching the schedule of the VN group.
  Interventions: Other: Basic Advice + Placebo Drug

INTERVENTIONS:
Other: Scheduled Gradual Reduction + Varenicline — Participants will receive a four-week Scheduled Gradual Reduction (SGR) intervention in which participants cut down on the number of cigarettes smoked. This is done through a smoking schedule in which participants smoke a cigarette at given fixed and equal intervals throughout their waking day. Additionally, they will take 0.5 mg of Varenicline (VN) once a day for the first three days, then 0.5 mg twice a day for the next four days, and they will continue for 13 weeks at 1.0 mg twice per day.
  Arms: Scheduled Gradual Reduction + Varenicline
Other: Scheduled Gradual Reduction + Placebo Drug — Participants will receive a four-week Scheduled Gradual Reduction (SGR) intervention in which participants cut down on the number of cigarettes smoked. This is done through a smoking schedule in which participants smoke a cigarette at given fixed and equal intervals throughout their waking day. Additionally, they will take placebo pills matching the schedule of the VN group.
  Arms: Scheduled Gradual Reduction + Placebo Drug
Other: Basic Advice + Varenicline — Participants will receive informational pamphlets with advice about quitting smoking. Additionally, they will take 0.5 mg of Varenicline (VN) once a day for the first three days, then 0.5 mg twice a day for the next four days, and they will continue for 13 weeks at 1.0 mg twice per day.
  Arms: Basic Advice + Varenicline
Other: Basic Advice + Placebo Drug — Participants will receive informational pamphlets with advice about quitting smoking. Additionally, they will take placebo pills matching the schedule of the VN group.
  Arms: Basic Advice + Placebo Drug

SUMMARY:
This study has three main aims. Aim 1: To provide initial data on the efficacy of combined Scheduled Gradual Reduction (SGR) and Varenicline (VN) for smoking cessation, by assessing abstinence and levels of smoking at 2 time points (4 and 12 weeks post quit). Aim 2: To explore the possibility that SGR+VN will be particularly efficacious among smokers with higher background levels of Cue Reactivity (CR), as assessed at the start of the study, using a classic experimental smoking CR paradigm. Aim 3: To explore possible mechanisms underlying the effects of SGR+VN, by assessing potential mediators (i.e., self-efficacy, cue-induced cravings) of treatment effects.

DETAILED DESCRIPTION:
Smoking remains an intransigent public health concern. There is ample evidence that non-pharmacological factors, such as environmental triggers (e.g., sight or smell of a cigarette), can give rise to strong classically-conditioned urges to smoke (termed 'cue-reactivity' [CR]), and that exposure to smoking cues can contribute to cessation failure. One promising intervention that may address CR is scheduled smoking with gradual reduction (SGR). Under SGR, individuals smoke only at fixed intervals, and over several weeks, systematically decrease their cigarettes consumed each day. The approach is postulated to: 1) provide 'practice' coping with environmentally-triggered cravings that occur during the inter-cigarette intervals, yielding increased self-efficacy to quit, and 2) weaken the associations between cues and smoking. Accumulating evidence has also shown that the smoking cessation drug, varenicline (VN), substantially ameliorates cravings and enhances cessation, significantly outperforming other drugs. Interestingly, recent animal research suggests that VN may operate at least partially by dampening conditioned drug cravings. A combination therapy consisting of SGR+VN might thus lead to significantly enhanced cessation, simultaneously attacking cravings using both pharmacological and non-pharmacological approaches. Because the beneficial effects of SGR and VN may be at least partially due to enhanced management of conditioned cravings, it is possible that that they will be particularly efficacious for smokers with high levels of CR. Using both laboratory experimental techniques and a prospective intervention design in this R34 application, we propose to provide initial data to: 1) test the hypothesis that a combination of SGR+VN will enhance cessation, 2) explore the possibility that SGR and VN might be particularly efficacious among smokers with higher levels of CR, and 3) explore potential mechanisms underlying treatment effects. Findings from this study would set the stage for larger efficacy and effectiveness trials of SGR alone and in conjunction with VN, as well as efforts to target SGR and/or VN toward the subgroups that would benefit the most (e.g., smokers with high levels of CR, carriers of specific smoking-related genotypes).

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker
* Averages at least 10 cigarettes/day for 5 or more years
* DSM-IV diagnosis of Nicotine Dependence
* Breath carbon monoxide > 6 ppm
* Motivated to quit: score > 8 on Contemplation Ladder
* Age > 18 years

Exclusion Criteria:

* Current illicit substance use
* Other tobacco use (e.g., cigar, pipe)
* History of psychosis
* Past or current cardiovascular disease
* Impaired renal functioning
* Pregnancy
* Nursing
* Current treatment for smoking cessation
* Clinically significant depressive symptoms (CES-D > 16)
* Current suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of Prolonged Abstinence | up to12 weeks post-quit
  Prolonged Abstinence from 12 weeks post-quit as compared to 4 weeks post-quit

SECONDARY OUTCOMES:
Comparison of Continuous Abstinence | 30 days post-quit and 30 days post end-of-treatment
  Continuous Abstinence as compared from 30 days post-quit to 30 days post end-of-treatment
Comparison of Survival | 30 days post-quit and 30 days post end-of-treatment
  Survival as compared from 30 days post-quit to 30 days post end-of-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joel Erblich, Ph.D, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273